CLINICAL TRIAL: NCT02429921
Title: Mitigating Arsenic Toxicity in Bangladeshi People by Supplementing Their Diets With High Selenium Lentils
Brief Title: High-selenium Lentils Versus Arsenic Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Judit E.G. Smits, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB13-1211_MOD1
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Arsenic Poisoning
Keywords: dietary intervention; arsenic poisoning; high-Se lentils
MeSH Terms: conditions — Arsenic Poisoning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-Se lentils (Experimental): 50 mg of low-selenium lentils per person consumed as soups
  Interventions: Dietary Supplement: Low-Se lentils
- high-Se lentils (Experimental): 50 mg of high-selenium lentils per person consumed as soup
  Interventions: Dietary Supplement: high-selenium lentils

INTERVENTIONS:
Dietary Supplement: high-selenium lentils — lentils grown on naturally selenium-rich soils in the Canadian Prairies
  Arms: high-Se lentils
Dietary Supplement: Low-Se lentils — lentils grown on selenium-deficient soils in Idaho, USA.
  Other Names: low-selenium lentils
  Arms: low-Se lentils

SUMMARY:
About 45 million people in Bangladesh are chronically exposed to unacceptable levels of arsenic in their drinking water. Chronic arsenic poisoning leads to cancers, and vascular diseases.

This dietary trial intends to test the potential of high-selenium lentils, consumed as lentil soup, in reducing the arsenic body burden in an exposed Bangladeshi population, and in improving the overall health status.

Arsenic-exposed families will be assigned to one of two groups. One group will eat lentils (50g/person/day) that are naturally high in selenium, the other group will receive lentils with low selenium content. This 6 months trial is randomized and double-blinded.

DETAILED DESCRIPTION:
Chronic arsenic (As) poisoning is a worldwide public health problem. Up to 100 million people worldwide, are chronically exposed to dangerously high concentrations of As in their drinking water and food supply. Bangladesh is facing a major public health challenge - contamination of groundwater by arsenic (As). Since tube well water contamination by As was discovered in Bangladesh in the 1990s, As in drinking water has been reduced by 40%, yet approximately 45 million Bangladeshis remain at risk from high As concentrations greater than the WHO guideline value of 10 µg/L in the well water. The annual cost to treat As related health problems in Bangladesh is currently estimated up to $77.5 million. Micronutrient-deficient (e.g. Selenium) soils lead to less nutritious local foods, which becomes a partner in crime exacerbating the toxic burden incurred by As exposure.

Selenium (Se) is a trace element that is an essential component of several metabolic pathways controlling immune function. Se and As work antagonistically in the body by competing in many biological functions. Arsenic added to animal diets has been known to counteract Se toxicity/activity in animals since the 1930s. Se interacts with As to form a complex; excessive Se excretion can occur as result of Se/As complex formation under condition of chronic As ingestion and low dietary Se ingestion. This scenario may further accelerate Se depletion. Again, since Se can form a complex with As, Se supplementation, in principle, can reduce As toxicity and also decrease effects of As exposure on many other parameters, such as oxidative stress, immunotoxicity etc.

Supplementation of Se as pills is currently used to treat arsenicosis. But pills are not often well received by people and are expensive for low-income families. Lentils are a common food in Bangladesh and the country already imports lentils from Canada. Saskatchewan (SK) grown lentils are rich in Se, mostly in form of L-selenomethionine, which is highly bioavailable. The Saskatchewan lentils have mean selenium levels between 425-672 µg/kg, with some regions where lentil selenium levels go up to 1884 µg/kg. These high Se lentils, incorporated into the daily meals of As-exposed Bangladeshi families, may help mitigate the symptoms of long-term As poisoning in a cost-effective, uncomplicated, and nutritionally beneficial way.

Red lentils for this trial were grown in Saskatchewan, Canada (Se = 854 µg/kg) and Idaho, USA (Se = 0.043 µg/kg). Other nutrients will be measured in both crops of lentils at the UofS before dispatching to families in Bangladesh. High-Se and low-Se lentils will be packed in two different coloured packets and will be given to the designated families. The investigators as well as the field staff will be blinded to the types of lentils/dahl being given to each family. 65g lentils per person/day will be measured with a cup by the female family head, who typically cooks the moshur dahl (lentil soup) daily for the whole family. 65g high-Se lentils provide 55 µg Se, which is the recommended daily allowance of 55 µg/person/day.

Sampling procedure and Data collection: At the start, at mid-term and the end of the trial (Table 1), household water samples, plus hair, blood, faeces and on-spot urine samples will be collected from each individual.

Water (20 ml): Currently used drinking water for measurement of arsenic, and other toxic and essential elements. Water will be acidified before storage at pH <2.0 in trace element free tubes at room temperature.

Urine (15-20 ml): Urine will be collected in trace element free tubes, aliquoted and stored in -80°C.

Stool (5-10 g): Stool will be collected in trace element free tubes and stored in -20°C.

Blood (5 ml/visit): Blood will be collected using a sterile needle and syringe in trace element free vacutainer tubes. Blood samples will be sent to Dhaka Lab on the same day in cool boxes and separated into plasma and cells, aliquot of plasma will be stored at -80°C. Buffycoat cells will be stored in RNALater in -80°C freezer. Whole blood (100 ul) will be stored in -80°C.

Hair: Hair from the back of the head will be collected (about 0.2 g) for analysis of As, as hair As is a suitable marker for long term exposure.

Laboratory Methods:

Metals: Se will be measured in blood by Graphite Furnace Atomic Absorption Spectrometry (GFAAS). Arsenic in hair, stool and urine samples will be measured by Hydride Generation Atomic Absorption Spectrometry (HGAAS) after acid digestion of samples.

Oxidative stress and antioxidant status : the investigators will measure 8-oxo-7, 8-dihydro-2'-deoxyguanosine (8-oxodG), a major product of ROS-induced oxidative stress, in urine/plasma of children using commercial ELISA kits. Reduced glutathione (GSH) is considered as an important scavenger of reactive oxygen species (ROS), and its ratio with oxidized glutathione (GSSG) is used as a marker of oxidative stress. The antioxidant status (GSH/GSSG) in whole blood will be assessed by measuring GSH and GSSG using commercial kits.

Lung inflammation: The investigators will measure fractional exhaled nitric oxide (FENO) in participants (≥9 yrs) as a marker of allergic lung inflammation. Monitoring FENO is simple and non-invasive with the use of a hand held small equipment. FENO will be measured online by the single breath technique according to published guidelines (ref) and manufacturer's instructions, with a NIOX MINO®. FENO will be recorded as mean value from two successive reproducible readouts. FENO data will be given as p.p.b. NIOX MINO uses IR communication for transfer of participant data to a PC using the software NIOX MINO Data Manager. FENO is usually high in individuals with current allergic asthma or rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* low, moderate and high arsenic levels in tube well water, that the household uses. If tube well water exceeds the national standard of 50 ppb, families will be advised to switch to another well in their proximity with lower Arsenic levels, if available.

Exclusion Criteria:

* Families that have very low arsenic levels (below US standard of 10 ppb) in their well water will not be enrolled.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
arsenic body burden | week 12
  Urine, feces, and hair samples of participants will be tested for arsenic content.

SECONDARY OUTCOMES:
Antioxidant status | week 24
  Blood specimen will be tested for glutathione (ox/red) levels.
oxidative damage | week 24
  Blood specimen will be tested for 8-OHdG, a marker for oxidative DNA damage.
serum lipid levels | week 24
  Serum will be analyzed for triglyceride, total cholesterol, HDL- and LDL-cholesterol.
Lung inflammation test | week 12
  Participants will exhale into a NIOX Mino device, which measures the nitric oxide level as marker of lung inflammation
Health and compliance questionnaires | biweekly (health) for 6 months
  Health questionnaire (and initial sociodemographic questionnaire) will be filled in by participant every two weeks to assess overall health, and lentil consumption will be assessed weekly.
Body mass index | week 24
  Examination by health professionals: Body mass index
Blood pressure | week 24
  Examination by health professionals: blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Judit EG Smits, DVM, PhD, Principal Investigator — University of Calgary, Calgary, Alberta, Canada; Albert Vandenberg, PhD, Study Director — University of Saskatchewan
Locations (1):
- Field Office, International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Background] Zeng H, Uthus EO, Combs GF Jr. Mechanistic aspects of the interaction between selenium and arsenic. J Inorg Biochem. 2005 Jun;99(6):1269-74. doi: 10.1016/j.jinorgbio.2005.03.006. PMID 15917080
- [Background] Gailer J, George GN, Pickering IJ, Prince RC, Younis HS, Winzerling JJ. Biliary excretion of [(GS)(2)AsSe](-) after intravenous injection of rabbits with arsenite and selenate. Chem Res Toxicol. 2002 Nov;15(11):1466-71. doi: 10.1021/tx025538s. PMID 12437338
- [Background] Thavarajah D, Vandenberg A, George GN, Pickering IJ. Chemical form of selenium in naturally selenium-rich lentils (Lens culinaris L.) from Saskatchewan. J Agric Food Chem. 2007 Sep 5;55(18):7337-41. doi: 10.1021/jf070681i. Epub 2007 Aug 9. PMID 17685630
- [Background] Thavarajah D, Ruszkowski J, Vandenberg A. High potential for selenium biofortification of lentils ( Lens culinaris L.). J Agric Food Chem. 2008 Nov 26;56(22):10747-53. doi: 10.1021/jf802307h. PMID 18954072
- [Background] Thavarajah, D., et al. (2011), 'A global survey of effects of genotype and environment on selenium concentration in lentils (Lens culinaris L.): Implications for nutritional fortification strategies', Food Chemistry, 125 (1), 72-76.
- [Derived] Krohn RM, Raqib R, Akhtar E, Vandenberg A, Smits JE. A high-selenium lentil dietary intervention in Bangladesh to counteract arsenic toxicity: study protocol for a randomized controlled trial. Trials. 2016 Apr 27;17(1):218. doi: 10.1186/s13063-016-1344-y. PMID 27121115
- See also: WHO: Arsenic: Fact Sheet No. 372, December 2012. 2012. — http://www.who.int/mediacentre/factsheets/fs372/en/